CLINICAL TRIAL: NCT06901492
Title: The Diagnostic Application of PSMA PET/MR in Patients with PSA <20 Ng/ml and Initial Negative Prostate Biopsy
Brief Title: The Diagnostic Application of PSMAPET/MR in Patients Undergoing Secondary Prostate Puncture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20250225-08
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: PSMA PET/CT; Prostate Cancer; MpMRI
Keywords: Prostate cancer; PSMA PET/CT; mpMRI; Prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PET+/mpMRI+ group (Experimental): Patients in this group will undergo 68Ga-PSMA PET/mpMRI imaging, and the results show positive findings on both PSMA PET and mpMRI. These patients will undergo prostate biopsy guided by PSMA PET/CT.
  Interventions: Diagnostic Test: Prostate biopsy guided by PSMA PET/CT
- PET+/mpMRI- group (Experimental): Patients in this group will undergo 68Ga-PSMA PET/mpMRI imaging, and the results show positive findings on PSMA PET and negative on mpMRI. These patients will undergo prostate biopsy guided by PSMA PET/CT.
  Interventions: Diagnostic Test: Prostate biopsy guided by PSMA PET/CT
- PET-/mpMRI+ group (Active Comparator): Patients in this group will undergo 68Ga-PSMA PET/mpMRI imaging, and the results show negative findings on PSMA PET and positive on mpMRI. These patients will undergo prostate biopsy guided by mpMRI and US.
  Interventions: Diagnostic Test: Prostate biopsy guided by mpMRI/US
- PET-/mpMRI- group (Placebo Comparator): Patients in this group will undergo 68Ga-PSMA PET/mpMRI imaging, and the results show negative findings on both PSMA PET and mpMRI. These patients will undergo systematic prostate biopsy.
  Interventions: Diagnostic Test: Systematic prostate biopsy

INTERVENTIONS:
Diagnostic Test: Prostate biopsy guided by PSMA PET/CT — The patient will undergo pelvic non-contrast CT imaging. After co-registration of the CT images with 68Ga-PSMA PET/CT data at corresponding anatomical levels, a percutaneous gluteal approach will be utilized for CT-guided prostate biopsy.
  Arms: PET+/mpMRI+ group; PET+/mpMRI- group
Diagnostic Test: Prostate biopsy guided by mpMRI/US — The patient will undergo transrectal ultrasound (TRUS) prostate scanning. After co-registration and precise image fusion of TRUS findings with multiparametric MRI (mpMRI) data, a transperineal percutaneous approach will be employed to perform TRUS-guided prostate biopsy.
  Arms: PET-/mpMRI+ group
Diagnostic Test: Systematic prostate biopsy — The patient will undergo systematic prostate biopsy under TRUS guidance.
  Arms: PET-/mpMRI- group

SUMMARY:
The present study is designed to explore the value of targeted puncture guided by PSMA PET/CT or mpMRI in the diagnosis of patients with low PSA and initial negative prostate biopsy

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 years, male;
2. Serum PSA level 4-20 ng/mL;
3. Serum PSA level 4-20 ng/mL;
4. No contraindications to PSMA-PET/CT or MRI;
5. Signed informed consent.

Exclusion Criteria:

1. Serum PSA >20 ng/mL;
2. History of prostate surgery/radiotherapy;
3. Acute prostatitis;
4. Coagulation disorders or active infection;
5. Severe internal/external hemorrhoids, perianal, rectal, or gluteal lesions;
6. Allergy to local anesthetics;
7. Inability to tolerate the biopsy procedure.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Biospy outcome | 12 months
  Compare the diagnostic value (including sensitivity, specificity, NPV and PPV) between puncture methods and set up a diagnostic model.

SECONDARY OUTCOMES:
Duration of puncture operation | 12 months
  Record the time required for each patient's puncture procedure
Patient's pain level | 12 months
  Based on VAS pain score
Blood loss | 12 months
  Bleeding volume during and after operation
Complication | 12 months
  Complications during and after the operation, including urethral injury, hematuria, and urinary tract infection, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No